CLINICAL TRIAL: NCT05200273
Title: A Phase 1a, Multicenter, Open-label, Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK114 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK114
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK114-102
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Advanced or Metastatic Solid Tumors; Malignancy; Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Non Randomised
Masking Description: None (open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): Experimental
  Interventions: Drug: AK114

INTERVENTIONS:
Drug: AK114 — AK114 administered by subcutaneous injection

SUMMARY:
A Phase 1 study to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary antitumor activity of AK114.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1a, multicenter, open-label, single-arm dose-escalation study of AK114 to evaluate the safety, tolerability, PK, pharmacodynamics, antitumor activity and immunogenicity in adult subjects with advanced or metastatic solid tumors. The study is comprised of dose escalation phase. Approximately 30 subjects will be treated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent
2. Age ≥ 18
3. Subjects must have histologically or cytologically confirmed advanced or metastatic solid tumor
4. Subject must have at least one measurable lesion according to RECIST v1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1
6. At the time of Day 1 of the study, subjects with central nervous system (CNS) metastases must have been treated
7. Available archived tumor tissue sample (block or a minimum of 10 unstained slides of formalin-fixed paraffin-embedded tissues) to allow for correlative biomarker studies
8. Subjects may opt to provide two fresh biopsy samples (pretreatment and on treatment), where clinically appropriate
9. Adequate organ function
10. Use acceptable method of contraception from screening, and must agree to continue for 120 days after the final dose of investigational product

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other monoclonal antibodies
2. History or concurrent gastrointestinal perforation, surgery and wound healing complications, hemorrhage events
3. Patients with clinically significant cardiovascular disease
4. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of investigational product administration
5. Active or prior documented autoimmune disease within the past 2 years
6. History of primary immunodeficiency
7. History of organ transplant or hematopoietic stem cell that requires use of immunosuppressive medications
8. Known allergy or reaction to any component of the investigational product formulation.
9. History of interstitial lung disease or noninfectious pneumonitis except for those induced by radiation therapies.
10. Prior treatment with canakinumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From the time of informed consent signed through to 90 days after last dose of study drug
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study drug, whether or not considered related to the study drug.
Number of participants with a Dose Limiting Toxicity (DLTs) | Within the first 28 days after receiving the first dose of study drug
  DLTs will be assessed as having a suspected relationship to study drug according to pre-specific criteria in the protocol.

SECONDARY OUTCOMES:
Serum pharmacokinetics (PK) | From first dose of treatment through to 90 days after end of treatment
  Serum concentrations of study drug in individual subjects at different time points after study drug administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drgu through to 90 days after end of treatment
  The immunogenicity of study drug will be assessed by summarizing the number of subjects who develop detectable ADAs.
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed complete response (CR) or confirmed partial response (PR), based on RECIST Version 1.1.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the number (%) of subjects with best of response of confirmed CR or PR, or stable disease (SD) according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Alex HL Wong, MMedSc, Study Director — Akeso
Locations (1):
- Ashford Cancer Centre, Kurralta Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No